CLINICAL TRIAL: NCT05401526
Title: Ability of Challenge With 5 cmH2O of Positive End-expiratory Pressure to Predict Fluid Responsiveness in Prone Position: An Observational Study
Brief Title: Fluid Responsiveness in Prone Position
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Emre Sertaç Bingül, Medical Doctor, Lecturer, Istanbul University
Other Study IDs: 2022/629
Record Dates: First submitted 2022-05-26; First posted 2022-06-02 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Anesthesia; Spine Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We are planning to measure hemodynamic parameters (Heart Rate, Mean Arterial Pressure, Stroke Volume Index, Stroke Volume Variation, and Pulse Pressure Variation) and ventilatory parameters at four times (T1, T2,T3, and T4) during spinal operation at prone position. First measurement (T1, First baseline) will be performed in the prone position after performing tracheal intubation and confirming hemodynamic stability (defined as mean arterial pressure <10% for 3 minutes). After the T1 measurement, additional 5 cmH2O PEEP (Positive end-expiratory pressure) will be applied for 30 seconds which will be called as "short term low PEEP challenge (SLPC)". At the end of the SLPC and prior to PEEP lowering, T2 measurement will be performed and recorded. After the T2 measurement, PEEP will be decreased to the initial value (5 cmH2O) and three minutes later, a second baseline (T3) measurement will be performed. Thereafter, 500 ml isotonic saline will be loaded in 10 minutes. T4 measurement will be performed again three minutes after volume loading. All of the measurements will be completed before surgery start and surgical stimulus. Patients exhibiting an increase in stroke volume index more than 15% after fluid loading (between T3 and T4) will be classified as volume responders. Absolute pulse pressure variation change due to SLPC, Absolute Stroke volume variation change due to SLPC, stroke volume index percentage change due to SLPC, and stroke volume index percentage change after fluid loading will be calculated and compared. Our aim is to observe if short term low PEEP challenge has the ability to predict fluid responsiveness better than pulse pressure variation and stroke volume variation for patients operated in prone position.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spine surgery in prone position
* Age≥ 18 years
* Elective surgery

Exclusion Criteria:

* American Society of Anesthesiology physical status over III
* Valvular heart disease
* Any ventricular dysfunction
* Preoperative arrythmias
* Preoperative hemodynamic instability
* Preoperative uncontrolled hypertension
* Preoperative uncontrolled diabetes mellitus
* History of lung disease
* Morbid obesity (Body mass index ≥ 40 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing spine surgery in prone position
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Verification of stroke volume index percentage change after SLPC | Up to 30 minutes
  Stroke volume index percentage change after SLPC means " [(SVIT2 - SVIT1) / SVIT1] x 100".
Verification of stroke volume index percentage change after fluid loading | Up to 30 minutes
  Stroke volume variation and pulse pressure variation values will be measured at second baseline (T3) and after fluid loading (T4).
  Fluid responsive patients means " stroke volume index increase after fluid loading ≥ 15%".
  In another explanation; [(SVIT4- SVIT3)/ SVI (T3)]x100 ≥ 15% means fluid responsive patients.
Ability of fluid responsiveness prediction with SVV, PPV, and Stroke volume index percentage change after SLPC | Up to 30 minutes
  Predictive ability of SVI changes after SLPC and fluid loading will be compared by statistical analysis (ROC curve)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ali A, Aygun E, Abdullah T, Bolsoy-Deveci S, Orhan-Sungur M, Canbaz M, Ozkan Akinci I. A challenge with 5 cmH2O of positive end-expiratory pressure predicts fluid responsiveness in neurosurgery patients with protective ventilation: an observational study. Minerva Anestesiol. 2019 Nov;85(11):1184-1192. doi: 10.23736/S0375-9393.19.13721-2. Epub 2019 Jun 17. PMID 31213047